CLINICAL TRIAL: NCT00703365
Title: A Multicenter, Open Label, Single Arm, Phase II Study to Investigate the Efficacy and Safety of Sorafenib (Nexavar) in Combination With Gemcitabine in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Efficacy and Safety of Sorafenib (Nexavar) in Combination With Gemcitabine in Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Bayer (Industry); Chulalongkorn University (Other); Bumrungrad International Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12849
Record Dates: First submitted 2008-05-20; First posted 2008-06-23 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sorafenib
  Interventions: Drug: Sorafenib and Gemcitabine

INTERVENTIONS:
Drug: Sorafenib and Gemcitabine — Sorafenib 400 mg po bid daily and Gemcitabine IV 1,000 mg/m2 on day 1,8, 15 of a 28-day cycle (up to 6 cycles), then followed by Sorafenib 400 mg po bid daily maintenance until disease progression.
  Other Names: Nexavar and Gemzar

SUMMARY:
This study is to evaluate the efficacy and safety of Sorafenib in combination with Gemcitabine in patients with advanced/unresectable HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), also known as primary liver cancer, is the fifth most common cancer in the world. It is responsible for about 90 percent of the primary malignant liver tumors observed in adult and disproportionately affects men, with about three times as many men developing the disease as women.

Common symptoms in patients affected with HCC include abdominal pain, weight loss, weakness, fullness and anorexia, abdominal swelling, jaundice and vomiting.

Multiple clinical staging systems for hepatic tumors have been used such as the American Joint Committee on Cancer TNM system (stage 0, A, B, C, D) etc. However, the staging systems are still evolving with all attempts to improve the classification and prognosis prediction of HCC, and there is no agreement on the best staging that can be recommended world-wide.

For advanced HCC, sorafenib is likely to become the new standard of care. Combinational therapies with sorafenib have the potential to further improved therapeutic options for patients suffering from advanced HCC. Gemcitabine is a classical chemotherapeutic substance that has modest anti-cancer activity in HCC. However, its anti-cancer activity seems to be improved when combined with other anti-cancer drugs including drugs interfering with the VEGF pathway. Both substances, sorafenib and gemcitabine, have a favorable safety profile with a minimal overlap of side effects. Further the mode of actions of sorafenib and gemcitabine are likely to result in synergistic anti-tumor effects.

An open label, single arm, multicenter phase II study designed to determine progression free survival of patients with advanced stage HCC treated with sorafenib in combination with gemcitabine. Patients will receive up to 6 cycles of gemcitabine(IV 1000 mg/m2 on day 1, 8, 15 of a 28-day cycle) in combination with sorafenib (400 mg po bid daily) followed by sorafenib (400 mg po bid daily) maintenance until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* patient at least 18 years of age with written informed consent prior to enrollment into the study.
* histologically or cytologically confirmed advanced unresectable and/or metastasis) HCC
* Child-Pugh class A or B
* Have measurable disease according to RECIST criteria
* life expectancy of at least 12 weeks, ECOG 0-2
* Have adequate bone marrow reserve and liver and renal function at screening
* Practice adequate contraception during study participation

Exclusion Criteria:

* Exclude medical conditions including history of cardiac disease, HIV infection,active infection,brain metastastasis or intracranial metastasis,seizure disorder requiring medication, history of organ allograft,evidence of or history of bleeding diathesis,previous or concurrent cancer with distinct in primary site or histology (with exception of cervical carcinoma in situ and treated basal cell carcinoma
* Excluded therapies and medications, previous and concomitant : prior systemic anticancer chemotherapy or immunotherapy or targeted therapy,hormonal therapy within 2 weeks,local treatment modality within 4 weeks,radiotherapy within 3 weeks,major surgery and unhealed wound within 4 weeks,autologous bone marrow transplant or stem cell rescue within 4 months
* other condition that may interfere with the patient's participation in the study or evaluation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (progression free survival (PFS)) of sorafenib in patients with advanced/unresectable HCC. | 2.5 years

SECONDARY OUTCOMES:
To evaluate overall, survival, overall response rate (RECIST), time to progression (TTP), disease control rate (DCR) and side-effect profile of sorafenib in combination with gemcitabine in patients suffering from HCC. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vichien Srimuninnimit, Assist.Prof., Principal Investigator — Siriraj Hospital, Bangkok, Thailand
Locations (3):
- Thailand (3):
  - Department of Medicine, Siriraj Hospital, Bangkoknoi, Bangkok
  - Medical Oncology Unit, Chulalongkorn Hospital, Patumwan, Bangkok
  - Horizon Regional Cancer Center, Bamrungrad Hospital, Sukhumvit, Bangkok

REFERENCES:
- [Background] Louafi S, Boige V, Ducreux M, Bonyhay L, Mansourbakht T, de Baere T, Asnacios A, Hannoun L, Poynard T, Taieb J. Gemcitabine plus oxaliplatin (GEMOX) in patients with advanced hepatocellular carcinoma (HCC): results of a phase II study. Cancer. 2007 Apr 1;109(7):1384-90. doi: 10.1002/cncr.22532. PMID 17330837